CLINICAL TRIAL: NCT02566356
Title: Mechanisms and Effects of Oxytocin on Social Cognition in Schizophrenia - fMRI
Brief Title: Adult Study Oxytocin - fMRI
Acronym: ASO-fMRI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joshua Woolley, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12-09654
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Schizophrenia; Oxytocin; Social Cognition; Functional Magnetic Resonance Imaging (fMRI)
Keywords: Oxytocin; Syntocinon; Social Cognition; Schizophrenia; Functional Magnetic Resonance Imaging (fMRI)
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): 40 IU Oxytocin
  Interventions: Drug: Oxytocin
- Saline Nasal Spray (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Saline Nasal Spray

INTERVENTIONS:
Drug: Oxytocin — 40 IU of the oxytocin will be administered intranasally for a one time dose at the beginning of the visit.
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Saline Nasal Spray — 40 IU of the saline nasal spray will be administered once at the beginning of the visit.
  Other Names: Placebo
  Arms: Saline Nasal Spray

SUMMARY:
In this study, investigators will examine the behavioral effects and neurophysiological mechanisms of the pro-social neuropeptide oxytocin in patients with recent-onset schizophrenia. Such research is a necessary first step towards identifying whether intranasal oxytocin administration can serve as an adjunct treatment for social impairments in schizophrenia.

Aim 1: To examine the effects of exogenous oxytocin on patterns of neural activation as measured by fMRI during a well-characterized affect-labeling task in patients with recent-onset schizophrenia and healthy comparison subjects.

Hypothesis A: Patients will exhibit amygdalar hyperactivity and PNS hypo-activity when passively viewing faces, which will be normalized by administration of oxytocin.

Hypothesis B: Patients will exhibit hypo-activity of the vPFC when affectively labeling faces and this hypo-activity will be normalized by oxytocin administration.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Male
* SCID-IV confirmed diagnosis of schizophrenia or schizoaffective disorder
* Clinically stable
* No changes to medications for the past week

Inclusion Criteria for Healthy Controls:

* Male
* SCID-IV confirmed no diagnosis of a current Axis I disorder within the last year

Exclusion Criteria for Patients and Healthy Controls:

* Meeting criteria for current substance abuse or dependence or illicit drug use within the last month (nicotine use is acceptable) as determined by a Urine Toxicology Drug Screening
* Any illness that affects the nasal passages and impairs the delivery of a nasal spray
* Presence of any neurological or significant medical disorder, including medical illnesses that could interfere with physiological recording such as cardiac arrhythmias
* A pacemaker, extensive dental work, or any magnetic metal implants and upper body tattoos
* Pregnancy
* Claustrophpbia
* Hearing difficulties
* A history of seizures
* Failure to receive a passing score on the reading test

Additional Exclusion Criteria for Patients and Healthy Controls:

* Taking any psychotropic medication or any medication that affects the autonomic or cardiovascular systems.
* Schizophrenia or other psychotic disorder in a first degree relative
* Failure to receive a passing score on the MOCA

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2012-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in fMRI neural activation patterns | 2-days at least 1-week apart
  During tasks in which participants will see and hear various stimuli, investigators will measure the change in neural activity in the medial prefrontal cortex and the temporoparietal junction between placebo and oxytocin testing days using the fMRI 3T Siemens Skyra scanner.

SECONDARY OUTCOMES:
Quality of Life Scale (QLS) | 1 day
  The QLS is a 21-item clinical rating scale where the interviewer rates the participant's responses on a scale of 1-6 where 6 indicates no impairment. In the fMRI study an abbreviated version of the QLS is used that includes 9 of the 21 items. The 9 items are each derived from the sections examining interpersonal relations, occupational role functioning, intrapsychic foundations, and common objects.
Social Functioning Scale (SFS) | 1 day
  The SFS is designed to assess a subject's social skills and performance, and to measure functions that are of importance for schizophrenic patients. It is a 79-item scale completed by the subject.
UCLA Loneliness Scale | 1 day
  The UCLA Loneliness Scale assesses the loneliness level of participants. It is a 20-item scale where responses are measured from O ("I often feel this way") to N ("I never feel this way").
Experiences in Close Relationships - Relationship Structures (ECR-RS) | 1 day
  The ECR is used to evaluate the construct of adult attachment. The scale involves 36 itemized statements split into four parts, each part referring to a different attachment figure. Participants rank each item using a 7-point likert scale.
Parental Bonding Instrument (PBI) | 1 day
  The PBI measures fundamental parenting styles as perceived the child. The questionnaire is retrospective in that it asks the adult participant to answer the questions based on how they remember their parents to be during up until they were 16 years old. The measure is completed for both mothers and fathers separately. There are 25 questions where half the questions are focused on how the parent cared for them and half are focused on how the parents protected them. A likert scale is used to measure responses where 1 is agree (i.e. very like) and 4 is disagree (i.e. very dislike).
Premorbid IQ test (AmNART) | 1 day
  The American National Adult Reading Test (AMNART) is an instrument used to estimate premorbid verbal IQ in adults. Participants are shown 45 words one at a time and are asked to read the word aloud. The scorer then writes 0 if the participant read the word incorrectly or 1 if the pronunciation is correct.
Childhood Trauma Questionnaire (CTQ) | 1 day
  The CTQ is a brief survey of 6 early traumatic experiences, including death, divorce, violence, sexual abuse, illness or other. The scale determines and assesses an individual's understanding of their childhood trauma, if applicable.
Emotional Quotient Scale (EQS) | 1 day
  The EQ is a 60-item self-report questionnaire that is designed to measure empathy in adults. Participants use a 4 item likert scale to record their responses (1=definitely agree, 4= definitely disagree).
Kinsey Scale | 1 day
  The Kinsey scale attempts to describe a person's sexual orientation using a scale from 0 (i.e. heterosexual) to 6 (i.e. homosexual).
Socioeconomic Status (SES) | 1 day
  This assess participants' socioeconomic status through their educational level and occupational level using a scale from 1 (i.e. professional, higher executive level) to 7 (i.e. less than 7 years of school, unskilled employee). This scale is also used for the participants' primary and secondary caretakers.

CONTACTS AND LOCATIONS:
Overall Officials: Josh D Woolley, MD/PhD, Principal Investigator — University of California San Francisco, San Francisco Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California